CLINICAL TRIAL: NCT00325949
Title: A Phase 3, Open-Label Period Followed By a Randomized, Double-Blind, Placebo-Controlled Study of the Analgesic Efficacy and Safety of Extended Release Hydrocodone/Acetaminophen (Vicodin® CR) Compared to Placebo in Subjects With Chronic Low Back Pain
Brief Title: A Study of Pain Relief in Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Earle Lockhart, MD, Abbott Laboratories
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M05-790
Record Dates: First submitted 2006-05-11; First posted 2006-05-15 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Acetaminophen; Hydrocodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- arm label (1) hydrocodone/acetaminophen extended release (Experimental)
  Interventions: Drug: Extended release hydrocodone and acetaminophen (Vicodin CR)
- arm label (2) hydrocodone/acetaminophen extended release (Experimental)
  Interventions: Drug: hydrocodone/acetaminophen extended release (Vicodin CR)
- Arm label (3) placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Extended release hydrocodone and acetaminophen (Vicodin CR) — 2 tablets BID
  Other Names: hydrocodone / acetaminophen extended release
  Arms: arm label (1) hydrocodone/acetaminophen extended release
Drug: hydrocodone/acetaminophen extended release (Vicodin CR) — 1 tablet BID
  Other Names: hydrocodone/acetaminophen extended release
  Arms: arm label (2) hydrocodone/acetaminophen extended release
Drug: placebo — 2 tablets BID
  Arms: Arm label (3) placebo

SUMMARY:
This is a study of the safety and pain-relieving ability of extended release hydrocodone and acetaminophen tablets in patients with moderate to severe low back pain

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ages 21-75 years
* If female, must be of non-child bearing potential or practicing birth control
* Has a history of chronic low back pain for at least 6 months
* Requires medication for the management of the chronic low back pain
* Has sufficient pain to justify the use of around-the-clock opioids

Exclusion Criteria:

* Is associated with any currently ongoing research study, or has previously participated in a Vicodin CR study
* Is allergic or has had a serious reaction to hydrocodone, other opioids, or acetaminophen
* Cannot discontinue pain medications, even for the short time prior to the study start
* Has any clinically significant illness or recent injury, or has any significant laboratory abnormality, or has recently had major surgery, or plans to have surgery
* Has a history of gastric bypass surgery or preexisting gastrointestinal narrowing, or history of diseases that may narrow the gastrointestinal tract
* Has a history of malnutrition or starvation
* Has a history of drug (licit or illicit) or alcohol abuse or addiction, or consumes more than 4 alcoholic drinks per day
* Has a history of a major depressive episode within the past 2 years, or requires treatment with certain drugs for depression, or has a history of major psychiatric disorder
* Is a pregnant or breastfeeding woman
* Is incapacitated, bedridden, or confined to a wheelchair
* Has initiated any new therapy or medication for chronic low back pain within 1 month of screening
* Has had surgery, certain types of low back procedures, injured, or received certain medications for chronic low back pain within a certain specified time frame
* Has back pain due to or associated with certain types of conditions
* Has other conditions that may cause pain, such as rheumatoid arthritis, gout, or fibromyalgia

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Actual)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Difference from randomization baseline to each subject's final assessment | 12 Weeks
  Pain intensity difference assessed by the Chronic Low Back Pain Intensity Score (100mm Visual Analog Scale)

SECONDARY OUTCOMES:
Time to withdrawal due to lack of efficacy during the Double-blind Maintenance Period
Pain Intensity Difference from randomization baseline to each scheduled assessment
Global Assessments of Study Drug and Back Pain Status
Roland-Morris Disability Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Rita Jain, M.D., Study Director — Abbott
Locations (63):
- United States (63):
  - Site Ref # / Investigator 2216, Hueytown, Alabama
  - Site Ref # / Investigator 2605, Phoenix, Arizona
  - Site Ref # / Investigator 1990, Phoenix, Arizona
  - Site Ref # / Investigator 1974, Tempe, Arizona
  - Site Ref # / Investigator 1977, Tucson, Arizona
  - Site Ref # / Investigator 1992, Buena Park, California
  - Site Ref # / Investigator 1993, Burbank, California
  - Site Ref # / Investigator 2219, Fair Oaks, California
  - Site Ref # / Investigator 1989, Los Gatos, California
  - Site Ref # / Investigator 2157, Denver, Colorado
  - Site Ref # / Investigator 1994, Trumbull, Connecticut
  - Site Ref # / Investigator 2208, Clearwater, Florida
  - Site Ref # / Investigator 2210, DeLand, Florida
  - Site Ref # / Investigator 2207, Hollywood, Florida
  - Site Ref # / Investigator 2204, Miami, Florida
  - Site Ref # / Investigator 2205, Miami, Florida
  - Site Ref # / Investigator 2214, Oldsmar, Florida
  - Site Ref # / Investigator 2135, Plantation, Florida
  - Site Ref # / Investigator 2134, West Palm Beach, Florida
  - Site Ref # / Investigator 1975, Atlanta, Georgia
  - Site Ref # / Investigator 1991, Decatur, Georgia
  - Site Ref # / Investigator 1985, Chicago, Illinois
  - Site Ref # / Investigator 1978, Evansville, Indiana
  - Site Ref # / Investigator 1988, West Des Moines, Iowa
  - Site Ref # / Investigator 2580, Prairie Village, Kansas
  - Site Ref # / Investigator 2209, Metairie, Louisiana
  - Site Ref # / Investigator 1976, Shreveport, Louisiana
  - Site Ref # / Investigator 2203, Pasadena, Maryland
  - Site Ref # / Investigator 2603, Brockton, Massachusetts
  - Site Ref # / Investigator 2156, Wellesley Hills, Massachusetts
  - Site Ref # / Investigator 3420, Biloxi, Mississippi
  - Site Ref # / Investigator 2556, Florissant, Missouri
  - Site Ref # / Investigator 1980, St Louis, Missouri
  - Site Ref # / Investigator 1982, Missoula, Montana
  - Site Ref # / Investigator 1986, Omaha, Nebraska
  - Site Ref # / Investigator 3421, Las Vegas, Nevada
  - Site Ref # / Investigator 2206, Las Vegas, Nevada
  - Site Ref # / Investigator 1973, New York, New York
  - Site Ref # / Investigator 2578, Williamsville, New York
  - Site Ref # / Investigator 1983, Raleigh, North Carolina
  - Site Ref # / Investigator 2606, Raleigh, North Carolina
  - Site Ref # / Investigator 5161, Winston-Salem, North Carolina
  - Site Ref # / Investigator 2218, Cincinnati, Ohio
  - Site Ref # / Investigator 1995, Cincinnati, Ohio
  - Site Ref # / Investigator 1987, Cincinnati, Ohio
  - Site Ref # / Investigator 2211, Oklahoma City, Oklahoma
  - Site Ref # / Investigator 2215, Downingtown, Pennsylvania
  - Site Ref # / Investigator 2579, Duncansville, Pennsylvania
  - Site Ref # / Investigator 2213, Mechanicsburg, Pennsylvania
  - Site Ref # / Investigator 2137, Cranston, Rhode Island
  - Site Ref # / Investigator 2221, Greer, South Carolina
  - Site Ref # / Investigator 1984, Cordova, Tennessee
  - Site Ref # / Investigator 2217, Austin, Texas
  - Site Ref # / Investigator 2607, Bulverde, Texas
  - Site Ref # / Investigator 2590, Dallas, Texas
  - Site Ref # / Investigator 2117, Killeen, Texas
  - Site Ref # / Investigator 2604, Nederland, Texas
  - Site Ref # / Investigator 1979, Richardson, Texas
  - Site Ref # / Investigator 2212, San Angelo, Texas
  - Site Ref # / Investigator 1981, San Antonio, Texas
  - Site Ref # / Investigator 2220, San Antonio, Texas
  - Site Ref # / Investigator 2608, San Antonio, Texas
  - Site Ref # / Investigator 2158, Virginia Beach, Virginia